CLINICAL TRIAL: NCT01525173
Title: A Safety and Efficacy Study of ALPHAGAN® P and LUMIGAN® in Subjects Previously Treated With Latanoprost for Glaucoma and Ocular Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GMA-LUM-11-019
Record Dates: First submitted 2012-01-31; First posted 2012-02-02 (Estimated); Results first posted 2013-12-04 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-10

CONDITIONS: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — Bimatoprost; Lubricant Eye Drops; Latanoprost; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ALPHAGAN® P and LUMIGAN® (Active Comparator): 1 drop of latanoprost 0.005% ophthalmic solution once daily in each eye as run-in therapy for 30 days followed by 1 drop of 0.1% brimonidine tartrate ophthalmic solution (ALPHAGAN® P) 3 times per day and 1 drop of 0.01% bimatoprost ophthalmic solution (LUMIGAN®) once per day for 12 weeks.
  Interventions: Drug: 0.1% brimonidine tartrate ophthalmic solution; Drug: 0.01% bimatoprost ophthalmic solution; Drug: latanoprost 0.005% ophthalmic solution
- LUMIGAN® Alone (Active Comparator): 1 drop of latanoprost 0.005% ophthalmic solution once daily in each eye as run-in therapy for 30 days followed by 1 drop of 0.2% hypromellose lubricant eye drops (used for masking purposes) 3 times per day and 1 drop of 0.01% bimatoprost ophthalmic solution (LUMIGAN®) once per day for 12 weeks.
  Interventions: Drug: 0.01% bimatoprost ophthalmic solution; Drug: 0.2% hypromellose lubricant eye drops; Drug: latanoprost 0.005% ophthalmic solution

INTERVENTIONS:
Drug: 0.1% brimonidine tartrate ophthalmic solution — 1 drop of 0.1% brimonidine tartrate ophthalmic solution 3 times per day for 12 weeks.
  Other Names: ALPHAGAN® P
  Arms: ALPHAGAN® P and LUMIGAN®
Drug: 0.01% bimatoprost ophthalmic solution — 1 drop of 0.01% bimatoprost ophthalmic solution once per day for 12 weeks.
  Other Names: LUMIGAN®
Drug: 0.2% hypromellose lubricant eye drops — 1 drop of 0.2% hypromellose lubricant eye drops 3 times per day for 12 weeks.
  Other Names: GenTeal ®
  Arms: LUMIGAN® Alone
Drug: latanoprost 0.005% ophthalmic solution — 1 drop of latanoprost 0.005% ophthalmic solution once daily as run-in therapy for 30 days only.

SUMMARY:
This study will evaluate the efficacy and safety of either bimatoprost 0.01% ophthalmic solution (Lumigan®) alone or bimatoprost 0.01% ophthalmic solution (Lumigan®) and brimonidine tartrate 0.1% ophthalmic solution (Alphagan® P) in combination in patients previously treated with latanoprost 0.005% ophthalmic solution monotherapy who require additional intraocular pressure (IOP) lowering medication.

ELIGIBILITY:
Inclusion Criteria:

* Ocular hypertension or glaucoma in at least 1 eye
* Visual acuity of 20/100 or better in both eyes

Exclusion Criteria:

* Corneal refractive laser surgery (LASIK, LASEK, PRK, RK) in the study eye(s)
* Intraocular or glaucoma surgery in the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2012-01; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Deerfield Beach, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ALPHAGAN® P and LUMIGAN® | LUMIGAN® Alone
Started | 70 | 67
Completed | 63 | 62
Not Completed | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ALPHAGAN® P and LUMIGAN® | LUMIGAN® Alone | Total
Number analyzed (Participants) | 70 | 67 | 137
Age Continuous [Mean (Standard Deviation); unit: Years] | 65.7 (11.87) | 61.1 (13.91) | 63.4 (13.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 33 | 64
  Male | 39 | 34 | 73

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Diurnal Intraocular Pressure (IOP)
Description: IOP is a measurement of the fluid pressure inside the eye. IOP was measured in the study eye, defined as the worse eye at Baseline. The mean diurnal IOP is the average of all the IOP measurements in the study eye taken at 8 AM, 10 AM and 4 PM at Baseline and at Week 12. A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 12
Population: Per protocol population included all qualified participants who completed three months of treatment.
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- ALPHAGAN® P and LUMIGAN®: 1 drop of 0.1% brimonidine tartrate ophthalmic solution (ALPHAGAN® P) 3 times per day and 1 drop of 0.01% bimatoprost ophthalmic solution (LUMIGAN®) once per day for 12 weeks.
- LUMIGAN® Alone: 1 drop of 0.2% hypromellose lubricant eye drops (used for masking purposes) 3 times per day and 1 drop of 0.01% bimatoprost ophthalmic solution (LUMIGAN®) once per day for 12 weeks.
Arm/Group | ALPHAGAN® P and LUMIGAN® | LUMIGAN® Alone
Number analyzed (Participants) | 61 | 59
mm Hg
  Baseline | 22.3 (2.22) | 22.2 (2.44)
  Change from Baseline at Week 12 | -4.7 (2.55) | -4.0 (3.23)

ADVERSE EVENTS:
Arm/Group | ALPHAGAN® P and LUMIGAN® | LUMIGAN® Alone
Serious Adverse Events (participants affected / at risk) | 1/70 | 2/67
Other Adverse Events (participants affected / at risk) | 4/70 | 0/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ALPHAGAN® P and LUMIGAN® (N=70) | LUMIGAN® Alone (N=67)
Prolonged hospitalization cardiac ischemia (Cardiac disorders) | 0 | 1
Exacerbation of depression disorder (Psychiatric disorders) | 0 | 1
Esophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ALPHAGAN® P and LUMIGAN® (N=70) | LUMIGAN® Alone (N=67)
Ocular hyperemia (Eye disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.